CLINICAL TRIAL: NCT03389399
Title: Pulmonary Physiology and Systemic Inflammatory Signature Investigations in Early Onset Pulmonary Events Associated With Brigatinib Use in Non-Small Cell Lung Cancer and Other Diseases
Brief Title: Pulmonary Physiology and Systemic Inflammatory in EO Pulmonary Events With Brigatinib Use in NSCLC and Other Diseases
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Criterium, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-0846.cc
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Brigatinib; Early Onset Pulmonary Events
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Brigatinib 90 mg QD or brigatinib 90 mg QD x 7 days: This is a single-arm study of patients who plan on starting brigatinib 90 mg QD or brigatinib 90 mg QD x 7 days to brigatinib 180 mg QD. Study procedures include PFTs, 6minute walk test, Modified Borg dyspnea scale (mBDS), and phlebotomy before participants commence brigatinib and on days 2 and 8 of brigatinib treatment. Participants that develop a peak reduction in DLCO of 20% or more from baseline whose DLCO does not return to their baseline level on day 8 may, at the discretion of the investigator, undergo repeated testing on a subsequent time point (e.g., day 15) for serial observation to ensure resolution of EOPE if that is the suspected cause of DLCO reduction.

SUMMARY:
To estimate the incidence of Early Onset Pulmonary Events (EOPEs), defined as the proportion of participants with a peak reduction in DLCO of 20% or greater after commencing brigatinib at 90mg QD.

DETAILED DESCRIPTION:
This is a single-arm study of patients who plan on starting brigatinib 90 mg QD or brigatinib 90 mg QD x 7 days to brigatinib 180 mg QD. Participants who enroll on this study protocol will either be taking brigatinib in the context of an ongoing clinical trial, or as part of standard of care treatment as licensed by FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form, indicating that he or she has been informed of all pertinent aspects of the study, including the potential risks, and is willingly participating.
2. Stated willingness and ability to comply with all scheduled visits and study procedures, and be available for the duration of the study.
3. Be a male or female aged ≥ 18.
4. Must plan on receiving brigatinib at a starting dose of 90 mg QD, regardless of whether they are receiving brigatinib as a part of clinical trial (if they meet eligibility criteria for given clinical trial) or outside of clinical trial as part of standard of care cancer treatment per the FDA license.
5. Suitable for treatment with brigatinib per either FDA labels, an acceptable clinical indication or within brigatinib clinical trials.
6. Participants must plan on taking Brigatinib as the only systemic cancer treatment. This means that participants cannot be receiving other targeted therapies, chemotherapies, or immunotherapies while on brigatinib (Exceptions: nonimmunosuppressive supportive cancer therapies such as bone targeting agents [e.g., denosumab], and anti-emetics are allowed).
7. Must have Hemoglobin (Hb) of ≥10 g/dL.
8. Recovered from clinically relevant toxicities (in the opinion of the investigator) related to prior anticancer therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v4.03) grade ≤2.
9. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
10. Must have clearly documented information of previously received systemic cancer treatments including chemotherapy, immunotherapy, small molecule tyrosine-kinase inhibitors (incl. ALK-targeted TKI) and stop date of most recent systemic therapy.

Exclusion Criteria:

1. Have baseline oxygen supplementation requirement (i.e., resting O2 sats on room air ≥ 90%).
2. Have history or presence of pulmonary interstitial disease or drug-related pneumonitis on CT imaging of chest performed within 28 days prior to starting brigatinib.
3. Have malabsorption syndrome or other GI illness that could affect oral absorption of the study drug in the opinion of the investigator.
4. Have had a blood transfusion within past 120 days.
5. Have received any small molecule inhibitors, including crizotinib, within 7 days of the first dose of Brigatinib (e.g., If first scheduled dose of brigatinib is on a Monday, May 1st, 2017 then last dose of the prior line of small molecule inhibitor must have been given BEFORE Monday, April 24, 2017).
6. Have received cytotoxic chemotherapy, investigational agents, or cytotoxic doses of radiation within 14 days of brigatinib, except SRS or stereotactic body radiosurgery to anatomic sites not involving lung tissue.
7. Have received immunotherapy within 28 days of first dose of brigatinib.
8. Be on corticosteroid within 48 hours prior to first dose of brigatinib.
9. Have uncontrolled, or active cardiac, pulmonary or hematologic disease that can affect interpretation of DLCO, specifically including, but not restricted to:

   1. Pulmonary interstitial disease or drug-related pneumonitis
   2. Symptomatic or poorly controlled congestive heart failure (CHF) within 6 months prior to first dose
   3. Symptomatic or poorly controlled pulmonary embolism within last 6 months
10. Have an ongoing or active infection. The requirement for intravenous (IV) antibiotics is considered active infection.
11. Have a known or suspected hypersensitivity to AP26113 or its excipients.
12. Have any condition or illness that, in the opinion of the investigator, would compromise participant safety or interfere with evaluation of the drug study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study. Brigatinib is not administered by this study. Instead, participants will receive brigatinib as part of an ongoing thereapeutic clinical trial or will be prescribed brigatinib, which is now an FDA-approved drug. Entry criteria for this study will focus on those suitable for this observational study. Any brigatinib-related safety procedure or follow-up will also be set forth by the FDA label or the relevant clinical trial that is administering brigatinib to the participant in this study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
To estimate the incidence of Early Onset Pulmonary Events (EOPEs) | 8 days
  EOPEs is defined as the proportion of participants with a peak reduction in Diffusion capacity in the Lung of Carbon monoxide (DLCO) of 20% or greater after commencing brigatinib at 90mg once daily QD.

CONTACTS AND LOCATIONS:
Overall Officials: Camidge Ross, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (4):
  - University of Colorado Denver, Aurora, Colorado
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern Harold C Simmons Comprehensive Cancer Center, Dallas, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No